CLINICAL TRIAL: NCT04009252
Title: Effect of Multimodal Patient Education With a Personalized 3D Printed Model in Patients With Severe Periarticular Ankle Fractures
Brief Title: Patient Education Using 3D Printed Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019
Record Dates: First submitted 2019-06-12; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Ankle Injuries; Fracture, Ankle
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 3D model to be printed and used as teaching tool to discuss injury with patient as well as its associated long-term outcomes and potential complications. The operative plan will also be reviewed with the patient using the model as well as post-operative course (ie rehabilitation)
  Interventions: Behavioral: 3D Model Education
- Control Group (No Intervention): The CT image will be shown to the patients along with teaching

INTERVENTIONS:
Behavioral: 3D Model Education — A 3D model of the patients ankle fracture will be printed and used as a teaching tool to discuss long-term outcomes and potential complications.
  Arms: Intervention Group

SUMMARY:
Complex high energy fractures of the lower extremity are life changing injuries and are known to be associated with poor functional outcome post operatively. The list of potential post-operative complications associated with these injuries is long, and the worst of these fractures can even be limb threatening. One of the most difficult and prevalent post-operative issues this patient population faces is chronic pain and its association to opioid addiction, which is currently an epidemic across North America. These individuals not only present with physical insult but psychological trauma as well, which also greatly affects these patients post-operatively. Properly educating the patient about their injury and the process that they will embark on can greatly empower the patient as they begin their journey of rehabilitation. This process can hopefully mute or silence some of these modifiable risk factors predisposing patients to poor functional outcomes and chronic pain. The investigators also hope to help them initiate/develop coping strategies to better overcome the many obstacles these patients face and to do so using 3D printing. 3D printed models have not only been demonstrated to be valuable in orthopaedics, when it comes to educating patients about their disease and associated interventions, but many other specialties as well; such as: cardiac surgery, urology, and general surgery. Literature suggest that often little is understood or retained by the patient following a patient consent with regards to their injury, potential complications, interventions to be undertaken, as well as the rehabilitation process to follow. By providing the patient with a 3D printed model of their fracture while educating them pre-/post-operatively, the investigators hope they will better understand the aforementioned, often forgotten points, indirectly yielding better overall patient satisfaction, patient outcomes and pain scores.

ELIGIBILITY:
Inclusion Criteria:

* periarticular injury involving the plafond, calcaneus or talus that requires open reduction and internal fixation
* Patient must have a completed CT scan as part of their pre-operative planning protocol

Exclusion Criteria:

* open fracture
* patient with known psychiatric history (depression, borderline personality disorder, bipolar etc)
* prior fracture fixation of the same ankle or foot
* diabetic neuropathy/Charcot foot
* dementia or other cognitive comorbidities (ie stroke etc)
* no primary address
* patient who were not independent mobilizers prior to injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal Outcomes Data Evaluation and Management Scale (MODEMS) Expectations Questionnaire (expectations) | Change between pre-operative and 3 months after the patients operation
  The expectations of a patient in regards to their ankle surgery, this questionnaire is on a Likert scale from 1 to 5 with 1 indicating a worse score.
Musculoskeletal Outcomes Data Evaluation and Management Scale (MODEMS) Expectations Questionnaire (satisfaction) | 3 months post-operative
  The satisfaction of a patient in regards to their ankle surgery, this questionnaire is on a Likert scale from 1 to 5 with 1 indicating a worse score.

SECONDARY OUTCOMES:
Visual Analogue Score (VAS) for Pain | Change between pre-operative to 6 months post-operative, this questionnaire is on a Likert scale from 1 to 5 with 1 indicating a worse score.
  Patient will indicate on a scale from 1 to 10 cm on how bad they feel their pain is with a score of 1 indicating no pain and 10 indicating extreme pain.
SF-12 | Change between pre-operative to 6 months post-operative
  Measure of quality of life
Foot and Ankle Ability Measure (FAAM) | Change between pre-operative to 6 months post-operative
  Measure of ankle specific function

CONTACTS AND LOCATIONS:
Overall Officials: Karl Lalonde, MD, Principal Investigator — Clinical Investigator